CLINICAL TRIAL: NCT06970132
Title: A Phase Ib/II, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SY-5933 Tablets in Combination With CT-707 Tablets in Patients With Advanced Solid Tumors Harboring KRAS p.G12C Mutation
Brief Title: Study of SY-5933 Plus CT-707 in Advanced Solid Tumors With KRAS p.G12C Mutation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-5933-II-01
Record Dates: First submitted 2025-04-27; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
Keywords: KRAS p.G12C Mutation
MeSH Terms: interventions — conteltinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ib/II study of SY-5933 and CT-707 combination (Experimental): In Phase Ib, six KRAS p.G12C mutation-positive patients will first receive 800 mg QD SY-5933 and 600 mg QD CT-707 for dose escalation. The dose of CT-707 may be adjusted based on safety, pharmacokinetic and efficacy data. 1-2 regimens will be selected for an expansion phase.
  The Phase II study will treat KRAS p.G12C mutation-positive patients with SY-5933 and CT-707 across four tumor types (NSCLC, colorectal cancer, pancreatic cancer, and other solid tumors) until disease progression or intolerable toxicity.
  Interventions: Drug: SY-5933; Drug: CT-707

INTERVENTIONS:
Drug: SY-5933 — KRAS p.G12C inhibitor
  Other Names: SY-5933 tablet
Drug: CT-707 — Focal Adhesion Kinase (FAK) inhibitor
  Other Names: CT-707 tablet; SY-707 tablet; Conteltinib

SUMMARY:
This Phase Ib/II, open-label, single-arm study evaluates the safety, tolerability, pharmacokinetics, and preliminary efficacy of SY-5933 tablets combined with CT-707 tablets in patients with advanced solid tumors harboring the KRAS p.G12C mutation. The Phase Ib includes a dose-escalation phase to determine the optimal dosing regimen based on safety and pharmacokinetic data. In Phase II, four cohorts will be enrolled: advanced KRAS p.G12C mutated non-small cell lung cancer (NSCLC), colorectal cancer, pancreatic cancer, and other solid tumors.

DETAILED DESCRIPTION:
This is an open-label, single-arm Phase Ib/II trial to assess the combination of SY-5933 and CT-707 in KRAS p.G12C mutated advanced solid tumors. In Phase Ib, six patients will receive 800 mg of SY-5933 and 600 mg of CT-707 once daily (QD) in a dose-escalation design, with dose adjustments based on safety, pharmacokinetic and efficacy data. The Ib expansion phase will further investigate the most promising dose/frequency combinations. In Phase II, four cohorts will be treated: advanced NSCLC, colorectal cancer, pancreatic cancer, and other solid tumors with KRAS p.G12Cmutation. Efficacy will be evaluated through interim analyses based on objective response rate. Patients will be treated until disease progression, unacceptable toxicity, death, or study completion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for enrollment in this study:

  1. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor.
  2. Age ≥ 18 years at the time of informed consent, regardless of gender.
  3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
  4. Life expectancy of at least 12 weeks.
  5. Presence of at least one extracranial target lesion (as defined by RECIST v1.1). Lesions previously treated with radiation therapy may only be considered target lesions if there is clear progression following radiation therapy.
  6. KRAS (G12C) mutation positive. For the Phase Ib dose-escalation phase, participants must have previously undergone standard treatment for advanced tumors. In the Phase II cohorts: Cohort 1 (NSCLC), Cohort 2 (colorectal cancer), Cohort 3 (pancreatic cancer), and Cohort 4 (other solid tumors). In the Phase Ib expansion phase, except for NSCLC, patients with other tumor types must have previously undergone standard treatment for advanced tumors. For Cohort 2-4 of Phase II, initial enrollment will prioritize patients who have received prior standard treatment, but frontline patients may be considered if sufficient efficacy and safety data are collected during Phase Ib or the Phase II study, following review by the Safety Monitoring Committee (SMC) to assess the benefit-risk ratio.
  7. Adequate organ function as defined below:

     1. Liver function:

        Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3× upper limit of normal (ULN), or ≤ 5× ULN if liver metastasis is present.

        Total bilirubin (TBIL) ≤ 1.5× ULN, or ≤ 3× ULN and direct bilirubin (DBIL) ≤ 1.5× ULN if liver metastasis or Gilbert's syndrome is present.
     2. Bone marrow function (No blood products, hematopoietic growth factors, or other treatments for hematological abnormalities within 7 days prior to dosing):

        Absolute neutrophil count (ANC) ≥ 1.5×10^9/L. Platelet count (PLT) ≥ 75×10^9/L. Hemoglobin (Hb) ≥ 90 g/L.
     3. Renal function:

        Creatinine clearance ≥ 50 mL/min.
     4. Coagulation function:

     Prothrombin time (PT) or International Normalized Ratio (INR) ≤ 1.5× ULN (except for subjects on anticoagulation therapy).
  8. For women of childbearing potential, a negative serum pregnancy test must be obtained within 7 days prior to the first dose. Male and female participants of childbearing potential must agree to use adequate contraception or remain abstinent during the study and for at least 3 months after the last dose of investigational drug.
  9. Able to swallow oral medications and comply with the study protocol and follow-up requirements.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from this study:

  1. For patients in the Ib expansion cohort and Phase II, the presence of known major oncogenic driver alterations other than KRAS G12C mutation, such as EGFR, ALK, ROS1, RET, NTRK, KRAS G12D, etc. (Patients with co-mutations may be considered for enrollment after discussion with the investigator).
  2. Prior treatment with a KRAS p.G12C inhibitor.
  3. Receipt of chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, or other anti-tumor therapies within 3 weeks prior to the first dose of study drug, except for the following:

     1. Nitrosoureas or mitomycin C administered within 6 weeks prior to the first dose;
     2. Oral fluoropyrimidines and small molecule targeted agents administered within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose.
  4. Receipt of any investigational agents or therapies not yet approved for marketing within 4 weeks prior to the first dose.
  5. Underwent major surgery involving major organs (excluding needle biopsy) or experienced significant trauma within 4 weeks prior to the first dose.
  6. Adverse events from prior anti-cancer therapies have not recovered to Grade ≤1 as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 (except for toxicities assessed by the investigator as posing no safety risk, such as alopecia and Grade 2 peripheral neuropathy).
  7. Presence of spinal cord compression, leptomeningeal metastasis, symptomatic brain metastases, or CNS disease requiring escalating doses of corticosteroids. Subjects with previously treated and stable CNS metastases are eligible if neurologic function is stable, no new neurologic deficits are observed on clinical examination, and there is no evidence of radiographic progression for at least 4 weeks prior to the first dose. If corticosteroids are required for CNS metastases, the dose must have been stable for at least 2 weeks prior to study entry.
  8. Active infection requiring systemic anti-infective therapy within 2 weeks prior to the first dose.
  9. Active hepatitis infection (defined as HBsAg positive with HBV-DNA ≥2000 IU/mL; or HCV antibody positive with HCV-RNA ≥1000 IU/mL), HIV infection, or active syphilis (both non-treponemal and treponemal tests positive) that remains uncontrolled despite appropriate treatment, as assessed by the investigator.
  10. Presence of other severe pulmonary conditions requiring systemic treatment, such as active tuberculosis, interstitial lung disease, etc., that may, in the opinion of the investigator, affect study results or place the subject at unacceptable risk.
  11. History or presence of severe cardiovascular or cerebrovascular diseases/abnormalities, including but not limited to:

      1. Significant arrhythmias or conduction abnormalities requiring clinical intervention (e.g., clinically significant ventricular arrhythmias, Grade II-III atrioventricular block);
      2. Resting QTc interval corrected by Fridericia's formula (QTcF) >470 msec for females or >450 msec for males (Subjects with suspected drug-induced QTcF prolongation may be enrolled after investigator assessment and correction with medication if deemed safe);
      3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade ≥3 cardiovascular or cerebrovascular events occurring within 6 months prior to the first dose;
      4. New York Heart Association (NYHA) Class ≥II heart failure or left ventricular ejection fraction (LVEF) <50%;
      5. Uncontrolled hypertension despite optimal medical therapy, defined as an average systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg based on at least three repeated measurements at intervals of at least 10 minutes.
  12. Use of strong CYP3A inhibitors or inducers within 1 week or 5 half-lives (whichever is longer) prior to the first dose or anticipated use during the study period (Refer to Section 15.6 of the clinical trial protocol for details).
  13. History of malignancies other than the tumor type under investigation, except for: Malignancies that have been cured and have not recurred within 2 years prior to enrollment; Completely resected basal cell or squamous cell carcinoma of the skin; Completely resected carcinoma in situ of any type.
  14. Presence of significant gastrointestinal diseases that may affect drug absorption, including but not limited to active ulcerative colitis, Crohn's disease, peptic ulcer disease, or prior major gastrointestinal surgery significantly affecting absorption, as assessed by the investigator.
  15. History of hypersensitivity to any components or excipients of the study drug.
  16. Presence of poorly controlled pleural effusion, ascites, or pericardial effusion after intervention (defined as rapid re-accumulation or symptomatic recurrence within 2 weeks post-drainage requiring further intervention).
  17. Poorly controlled diabetes mellitus [defined as fasting blood glucose ≥10 mmol/L and/or HbA1c ≥8%], uncontrolled symptomatic hyperthyroidism or hypothyroidism, or uncontrolled symptomatic hypercalcemia or hypocalcemia.
  18. Coagulation disorders or bleeding diathesis, including but not limited to: History of arterial or venous thromboembolism within 6 months prior to the first dose (e.g., myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other serious thromboembolic events); History of life-threatening bleeding events (requiring transfusion, surgical or local intervention, or sustained medical treatment); Tumor invasion of major blood vessels posing a high risk of bleeding, as assessed by the investigator.
  19. Pregnancy or lactation.
  20. Any condition that, in the opinion of the investigator, may increase the risk associated with study drug administration, interfere with study results interpretation, affect subject compliance, or otherwise make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) in KRAS p.G12C Mutant Advanced Solid Tumors in Phase Ib | Up to 24 months
  Evaluate the safety and tolerability of SY-5933 combined with CT-707
Dose-limiting toxicity (DLT) of SY-5933 combined with CT-707 in KRAS p.G12C Mutant Advanced Solid Tumors in Phase Ib | From first dose to end of DLT observation period (approximately 28 days)
  To determine the recommended phase 2 dose (RP2D)
Objective response rate (ORR) of SY-5933 combined with CT-707 in KRAS p.G12C Mutant Advanced Solid Tumors in Phase II | Up to 24 months
  Evaluate the ORR based on RECIST v1.1 criteria to assess the preliminary efficacy of SY-5933 combined with CT-707 in patients with advanced solid tumors harboring KRAS p.G12C mutation

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | rotocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as maximum observed plasma concentration of investigational drugs
Pharmacokinetics (Tmax) | rotocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as time to maximum plasma concentration of investigational drugs
Pharmacokinetics (AUC0-t) | rotocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration of investigational drugs
Pharmacokinetics (t½) | rotocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as the apparent plasma terminal phase disposition half-life of investigational drugs
ORR of SY-5933 combined with CT-707 in KRAS p.G12C mutant advanced solid tumors in Phase Ib | Up to 24 months
  Evaluate the ORR based on RECIST v1.1 criteria to assess the preliminary efficacy of SY-5933 combined with CT-707 in patients with advanced solid tumors harboring KRAS p.G12C mutation
Incidence of adverse events (AEs) and serious adverse events (SAEs) in KRAS p.G12C mutant advanced solid tumors in Phase II | Up to 24 months
  Evaluate the safety and tolerability of SY-5933 combined with CT-707
Disease control rate (DCR) in Phase Ib and Phase II | Up to 24 months
  Evaluate the DCR based on RECIST v1.1 criteria to assess the preliminary efficacy of SY-5933 combined with CT-707 in patients with advanced solid tumors harboring KRAS p.G12C mutation
Duration of response (DoR) in Phase Ib and Phase II | Up to 24 months
  Evaluate the DoR based on RECIST v1.1 criteria to assess the preliminary efficacy of SY-5933 combined with CT-707 in patients with advanced solid tumors harboring KRAS p.G12C mutation
Progression-free survival (PFS) in Phase Ib and Phase II | Up to 24 months
  Evaluate the PFS based on RECIST v1.1 criteria to assess the preliminary efficacy of SY-5933 combined with CT-707 in patients with advanced solid tumors harboring KRAS p.G12C mutation

OTHER OUTCOMES:
Effect of SY-5933 combined with CT-707 on QT Interval Corrected by Fridericia (QTcF) | Up to 24 months
  Explore the effects of SY-5933 combined with CT-707 on QTcF and evaluate the relationship between plasma drug concentrations and QTcF interval changes
Baseline tumor FAK protein expression intensity | Up to 24 months
  Quantification of total FAK protein level in baseline tumor tissue via immunohistochemistry
Plasma phospho-FAK (Tyr397) levels | Up to 24 months
  Longitudinal measurement of phospho-FAK (Tyr397) Levels in peripheral blood using phospho-specific ELISA at baseline, first radiographic response assessment, and confirmed PD
Longitudinal plasma KRAS ctDNA variant allele frequency | Up to 24 months
  Dynamic quantification of KRAS p.G12C mutant burden in cell-free DNA via next-generation sequencing at baseline, first radiographic response assessment, and confirmed PD

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China